CLINICAL TRIAL: NCT06806319
Title: Soft Tissue Crown Lengthening and Attached Gingiva Remodeling: Assessment of Growth Factors Levels Associated with Wound Healing
Brief Title: Assessment of Growth Factors Levels Associated with Wound Healing After Soft Tissue Crown Lengthening
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: crown lengthening and gingiva
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Gingival Overgrowth
Keywords: Diode Laser; Electrosurgery; Crown Lengthening; Gingival crevicular fluid; Fibroblast Growth Factor; Platelet-Derived Growth Factor; Transforming Growth Factor beta1
MeSH Terms: conditions — Gingival Overgrowth; Hyperthermia; Camurati-Engelmann Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser crown lengthening technique (Active Comparator): 1-The patients were anesthetized using infiltration technique and/ or nerve block. 2-Specific protective glasses were used for patient, dentist, and assistant. Highly reflective instruments or instruments with mirrored surface were voided as there could be reflection of the laser beam. 3- The pocket depths in the surgical site were measured. Dots made in the gingiva by using Krane Kaplen tweezer, then area to be cut outlined by connection of dots (fig.6(D)) using Sirolase ® lower power diode laser 970 ± 15 nm (0.5 watts) continuous emission, power =3 watts, fiber 320 μm (fig.8). 4-Continue to split the dots halfway until there was a continuing line of dots by using the diode laser, 5-During the entire procedure, the tip was constantly checked for any debris of the ablated tissues and was cleaned with sterile moist gauze.6-Physiological gingival contour was achieved by changing the angulation of the tip as required during the procedure. 7-After the surgery, the end of the fiber (2-3mm)
  Interventions: Device: single intervention by Sirolase ® lower power diode laser 970 ± 15 nm (0.5 watts) continuous emission, power =3 watts, fiber 320 μm
- Electrocautery crown lengthening (Active Comparator): 1-Patients were anesthetized by infiltration technique and/ or nerve block 2-The pocket depths in the surgical site were measured using crane Kaplan tweezer. 3-Patient asked to hold the reusable silicone patient plate. 4-The output power of electrosurgical unit (fig.6) was kept 38 watts rms ± 5%. The working frequency was adjusted to 1.5 MHz ± 5%. 5-Continue to split the dots halfway until there was a continuing line of dots. 6-Avoid the operation of equipment in a room with flammable or explosive materials. 7-Rapid, well-planned movements without pressure and it should be like brushing strokes keep electrode moving all the time, use high enough current. 8-A cooling period of 8 seconds should be allowed between successive incisions with the electrode. 9-Continuous saline irrigation was given while using the electrocautery. 10-The excised tissues are removed with Orban knife.
  Interventions: Device: single intervention by electrosurgical unit which was kept 38 watts rms ± 5%. The working frequency was adjusted to 1.5 MHz ± 5%.

INTERVENTIONS:
Device: single intervention by Sirolase ® lower power diode laser 970 ± 15 nm (0.5 watts) continuous emission, power =3 watts, fiber 320 μm — single intervention by Sirolase ® lower power diode laser 970 ± 15 nm (0.5 watts) continuous emission, power =3 watts, fiber 320 μm.single intervention the follow-up until 6 months
  Arms: Laser crown lengthening technique
Device: single intervention by electrosurgical unit which was kept 38 watts rms ± 5%. The working frequency was adjusted to 1.5 MHz ± 5%. — single intervention by electrosurgical unit which was kept 38 watts rms ± 5%. The working frequency was adjusted to 1.5 MHz ± 5%.single intervention then follow-up until 6 months
  Arms: Electrocautery crown lengthening

SUMMARY:
Clinicians often encounter the need for crown lengthening in the practice of dentistry and have to make treatment decisions taking into consideration how to best address the biological, functional, and esthetic requirements of each particular case. The concept of crown lengthening was first introduced by D.W. Cohen (1962) and is presently a procedure that often employs some combination of tissue reduction or removal , osseous surgery , and/or orthodontics for tooth exposure and increasing the extent of supra gingival tooth structure for restoration of aesthetic purposes . Gingivectomy and gingivoplasty considered kind of crown lengthening procedure. Gingivectomy is defined as the excision of the soft tissue wall of a pocket. The procedure is usually combined with the recontouring of hyperplastic tissue by gingivectoplasty to restore physiological gingival form . Gingivoplasty is a reshaping of the gingiva to create physiologic gingival contours, with the sole purpose of recontouring the gingiva in the absence of pockets. In doing so, the complete anatomical crown becomes exposed and pseudo pockets are eliminated creating a better environment for periodontal health. Treatment options for crown lengthening procedures include: Surgical, Electrocautery or by Laser. The aim of the present study was to compare the practical effectiveness and postoperative parameters of using diode laser and electrocautery for crown lengthening procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 18 years. 2. Patients with short clinical crowns to enhance esthetic, exposure of subgingival caries for prosthetic replacement, exposure of a fracture or combination. 3. All patients were free from any systemic diseases according to the criteria of Modified Cornell Medical Index. 4. All patients need soft tissue removal and don't need osseous resection. 5. Full-Mouth Plaque Score (FMPS) ≤ 20% at baseline. 6. Full-Mouth Bleeding Score (FMBS) ≤ 20% at baseline.

Exclusion Criteria:

1. Light smokers i.e. smoking > 10 cigarettes/day. 2. Patients with medical conditions contraindicating surgical interventions. 3. Pregnancy or lactation. 4. Patients with active periodontal disease (PD ≥ 6 mm) 5. Clinical and/or radiographic signs of periapical pathology. 6. Patients with pacemakers.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Epithelization rate | From enrollment to the end of treatment at 3 weeks
  After gingivectomy operation, the surgical site was evaluated with hydrogen peroxide to detect the presence of epithelization. The mesio-distal width of the maxillary right central tooth was recorded for each patient, and photographs were calibrated via the reference values. all photographs were examined with the assistance of Image processing and analysis in Java, Image J software. In the areas subjected to hydrogen peroxide application and experiencing tissue reaction, there was a lack of an epithelial layer in the wound area.
Transforming Growth Factor-β1 (TGF-β1) levels assessment | From enrollment to the end of treatment at 8 weeks
  The levels of TGF-β1 in the GCF samples were determined using commercially available ELISA Kits

CONTACTS AND LOCATIONS:
Overall Officials: Asem M lecturer, PhD, Principal Investigator — Faculty of Dental Medicine, Al-Azhar University (Assiut branch)
Locations (1):
- Faculty of dental medicine, Al-Azhar University (Assiut branch), Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeballos BK, Rubina YN, Meza-Mauricio J, Cafferata EA, Vergara-Buenaventura A. Laser gingivectomy for maintaining periodontal health in fixed orthodontic patients: a systematic review. Lasers in Dental Science. 2024 Dec;8(1):1-5.
- [Background] Mehrotra S, Ahuja A, Chowdhary Z, Adhupia KS, Bajaj A, Loitongbam M. Evaluation of the Effect of Diode Laser on Healing after Gingivectomy. Pesquisa Brasileira em Odontopediatria e Clínica Integrada. 2025 Jan 15;25:e230116-.
- [Background] Rakmanee T, Calciolari E, Olsen I, Darbar U, Griffiths GS, Petrie A, Donos N. Expression of growth mediators in the gingival crevicular fluid of patients with aggressive periodontitis undergoing periodontal surgery. Clin Oral Investig. 2019 Aug;23(8):3307-3318. doi: 10.1007/s00784-018-2752-z. Epub 2018 Nov 29. PMID 30498980
- [Background] Kuru L, Yilmaz S, Kuru B, Kose KN, Noyan U. Expression of growth factors in the gingival crevice fluid of patients with phenytoin-induced gingival enlargement. Arch Oral Biol. 2004 Nov;49(11):945-50. doi: 10.1016/j.archoralbio.2004.04.010. PMID 15353252
- [Background] Guler B, Isler SC, Uraz A, Bozkaya S, Cetiner FD. The comparison of postoperative wound healing following different gingivectomy techniques: A randomized prospective clinical trial.